CLINICAL TRIAL: NCT05137925
Title: Exploring Mechanisms of Change in a Pilot Randomized Trial of Mindfulness-Based Cognitive Therapy to Promote Well-being During Pregnancy and Postpartum Among At-risk Pregnant Women
Brief Title: Mindful Moms: Mechanisms of Mindfulness-based Cognitive Therapy During Pregnancy and Postpartum
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: American Psychological Foundation (Other); The Pittsburgh Foundation (Other)
Responsible Party: Principal Investigator, Michele Levine, Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY21060191
Record Dates: First submitted 2021-10-26; First posted 2021-11-30 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Psychological Distress; Pregnancy Related; Postpartum Blues; Postpartum Depression; Postpartum Anxiety; Postpartum Sadness
MeSH Terms: conditions — Depression, Postpartum | interventions — Mindfulness-Based Cognitive Therapy; Therapeutics

STUDY DESIGN:
Intervention Model Description: The proposed study will randomize participants to an eight-week virtual group-based Mindfulness-based Cognitive Therapy intervention or to a treatment as usual control condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-Based Cognitive Therapy (MBCT) (Experimental): MBCT will be delivered in a group based, videoconference format with 90 minute sessions 1x/week.
  Interventions: Behavioral: Mindfulness-Based Cognitive Therapy (MBCT)
- Treatment as Usual (TAU) (Active Comparator): TAU, or the control group, provides information about the benefits of mindfulness in pregnancy, offers referrals for psychotherapy in the community, and involves monthly phone or videoconference calls to maintain engagement.
  Interventions: Behavioral: Treatment as Usual (TAU)

INTERVENTIONS:
Behavioral: Mindfulness-Based Cognitive Therapy (MBCT) — MBCT is an 8-week group-based treatment modality designed specifically to prevent recurrence of depressive symptoms. MBCT combines principles of cognitive behavioral therapy and mindfulness meditation to help participants change the way in which they relate to automatic negative thinking patterns that trigger symptom recurrence. Through awareness and acceptance of negative thoughts and emotions, participants learn how to dismiss negative thoughts and to tolerate distress and uncertainty.
  Arms: Mindfulness-Based Cognitive Therapy (MBCT)
Behavioral: Treatment as Usual (TAU) — TAU (the control group) provides participants with information about the benefits of mindfulness in pregnancy and offers referrals for psychotherapy in the community. Participants in TAU are contacted monthly via phone or videoconference call to maintain engagement.
  Arms: Treatment as Usual (TAU)

SUMMARY:
The proposed study seeks to elucidate the mechanisms underlying Mindfulness-Based Cognitive Therapy in pregnancy to improve understanding of how and why this treatment modality enhances well-being, which can then be leveraged to optimize treatment for psychological distress emerging during this vulnerable period.

DETAILED DESCRIPTION:
Pregnancy and postpartum is a period of vulnerability for new or worsening psychiatric symptoms. Mindfulness Based Cognitive Therapy (MBCT) is an effective approach to mitigate pregnancy-related worsening of psychological distress. However, prior research has focused predominantly on symptoms of depression and anxiety, and is it not clear how or why MBCT improves psychological health during the perinatal period. Thus, the goals of this project are to (1) examine whether MBCT improves psychological functioning among pregnant women and whether these improvements persist at three-months postpartum, (2) examine whether improved ability to regulate emotions and behavior accounts for the beneficial effects of MBCT, and (3) determine what demographic, socioeconomic, and psychosocial factors impact treatment engagement and effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* pregnancy between 12 and 30 weeks gestation
* reporting at least mild psychological distress (based on self-report)
* access to high-speed internet or cellular network access
* located in the U.S.

Exclusion Criteria:

* current suicidal or homicidal ideation as assessed verbally during screening
* symptom severity necessitating a higher level of clinical care
* current psychosis
* untreated mania
* active substance abuse
* lack of high-speed internet connection or cellular network access
* planning to be traveling without access to internet for more than two weeks in the next 12 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Change in presence and severity of depressive symptoms from baseline to 8 weeks | baseline and 8 weeks
  Change in the presence and severity of depressive symptoms from baseline to 8 weeks will be measured using the 10-item Edinburgh Postnatal Depression Scale (EPDS), a widely used instrument validated in pregnancy and the postpartum period. Questions 1, 2, 3, and 4 on the EPDS are scored 0, 1, 2, or 3 with the top box scored as 0 and the bottom box scored as 3. Questions 3 and 5-10 on the EPDS are reverse scored with the top box scored as 3 and the bottom box scored as 0. Total scores on the EPDS are calculated by summing the score for each question. Total scores on the EPDS range from 0-30, with a score of 10 or greater indicating possible depression and higher scores indicating greater severity of possible depression.
Change in presence and severity of depressive symptoms from 8 weeks to 3 months | 8 weeks and 3 months
  Change in the presence and severity of depressive symptoms from baseline to 3 months will be measured using the 10-item Edinburgh Postnatal Depression Scale (EPDS), a widely used instrument validated in pregnancy and the postpartum period. Questions 1, 2, 3, and 4 on the EPDS are scored 0, 1, 2, or 3 with the top box scored as 0 and the bottom box scored as 3. Questions 3 and 5-10 on the EPDS are reverse scored with the top box scored as 3 and the bottom box scored as 0. Total scores on the EPDS are calculated by summing the score for each question. Total scores on the EPDS range from 0-30, with a score of 10 or greater indicating possible depression and higher scores indicating greater severity of possible depression.
Change in perceptions of daily life stress from baseline to 8 weeks | baseline and 8 weeks
  Change in the perceptions of daily life stress from baseline to 8 weeks will be measured using the 10-item Perceived Stress Scale (PSS). Questions 1, 2, 3, 6, 9, and 10 on the PSS are scored 0, 1, 2, and 3. Questions 4, 5, 7, and 8 on the PSS are reverse scored 3, 2, 1, and 0. Total scores on the PSS are calculated by summing the score for each question. Total scores on the PSS range from 0-40, with higher scores indicating higher perceived stress. Scores ranging from 0-13 would be considered low stress, scores ranging from 14-26 would be considered moderate stress, and scores ranging from 27-40 would be considered high perceived stress.
Change in perceptions of daily life stress from 8 weeks to 3 months | 8 weeks and 3 months
  Change in the perceptions of daily life stress from 8 weeks to 3 months will be measured using the 10-item Perceived Stress Scale (PSS). Questions 1, 2, 3, 6, 9, and 10 on the PSS are scored 0, 1, 2, and 3. Questions 4, 5, 7, and 8 on the PSS are reverse scored 3, 2, 1, and 0. Total scores on the PSS are calculated by summing the score for each question. Total scores on the PSS range from 0-40, with higher scores indicating higher perceived stress. Scores ranging from 0-13 would be considered low stress, scores ranging from 14-26 would be considered moderate stress, and scores ranging from 27-40 would be considered high perceived stress.
Change in anxiety symptoms from baseline to 8 weeks | baseline and 8 weeks
  Change in anxiety symptoms from baseline to 8 weeks will be measured using the 16-item Penn State Worry Questionnaire (PSWQ). Questions 2, 4-7, 9, and 12-16 on the PSWQ are scored 1-5. Questions 1, 3, 8, 10, and 11 on the PSWQ are reverse scored 5-1. Total scores on the PSWQ are calculated by summing the score for each question. Total scores on the PSWQ range from 16-80, with higher scores indicating higher worry. Scores ranging from 16-39 would be considered low worry, scores ranging from 40-59 would be considered moderate worry, and scores ranging from 60-80 would be considered high worry.
Change in anxiety symptoms from 8 weeks to 3 months | 8 weeks and 3 months
  Change in anxiety symptoms from 8 weeks to 3 months will be measured using the 16-item Penn State Worry Questionnaire (PSWQ). Questions 2, 4-7, 9, and 12-16 on the PSWQ are scored 1-5. Questions 1, 3, 8, 10, and 11 on the PSWQ are reverse scored 5-1. Total scores on the PSWQ are calculated by summing the score for each question. Total scores on the PSWQ range from 16-80, with higher scores indicating higher worry. Scores ranging from 16-39 would be considered low worry, scores ranging from 40-59 would be considered moderate worry, and scores ranging from 60-80 would be considered high worry.
Change in rumination from baseline to 8 weeks | baseline and 8 weeks
  Change in rumination from baseline to 8 weeks will be measured using the 10-item Ruminative Response Scale (RRS-10). Questions 1-10 on the RRS-10 are scored 1-4. Total scores on the RRS-10 are calculated by summing the score for each question. Total scores on the RRS-10 range from 1-40, with higher scores indicating higher rumination.
Change in rumination from 8 weeks to 3 months | 8 weeks and 3 months
  Change in rumination from 8 weeks to 3 months will be measured using the 10-item Ruminative Response Scale (RRS-10). Questions 1-10 on the RRS-10 are scored 1-4. Total scores on the RRS-10 are calculated by summing the score for each question. Total scores on the RRS-10 range from 1-40, with higher scores indicating higher rumination.
Change in mindfulness from baseline to 8 weeks | baseline and 8 weeks
  Change in mindfulness from baseline to 8 weeks will be measured using the 39-item Five Facet Mindfulness Questionnaire (FFMQ). The FFMQ consists of five subscales, which are calculated by summing the following questions, which are scored 1-5 (questions followed by "R" are reverse scored 5-1): observing = questions 1, 6, 11, 15, 20, 26, 31, and 36; describing = 2, 7, 12R, 16R, 22R, 27, 32, and 37; acting with awareness = 5R, 8R, 13R, 18R, 23R, 28R, 34R, and 38R; nonjudging of inner experience = 3R, 10R, 14R, 17R, 25R, 30R, 35R, and 39R; nonreactivity to inner experience = 4, 9, 19, 21, 24, 29, and 33. For the FFMQ subscales, scores can range from 8 to 40, except for non-reactivity to inner experience, which can range from 7 to 35. For the FFMQ subscales, higher scores represent higher subscale levels of mindfulness. Total scores are calculated by summing the subscale scores and range from 39-195, with higher scores indicating higher overall levels of mindfulness.
Change in mindfulness from 8 weeks to 3 months | 8 weeks and 3 months
  Change in mindfulness from 8 weeks to 3 months will be measured using the 39-item Five Facet Mindfulness Questionnaire (FFMQ). The FFMQ consists of five subscales, which are calculated by summing the following questions, which are scored 1-5 (questions followed by "R" are reverse scored 5-1): observing = questions 1, 6, 11, 15, 20, 26, 31, and 36; describing = 2, 7, 12R, 16R, 22R, 27, 32, and 37; acting with awareness = 5R, 8R, 13R, 18R, 23R, 28R, 34R, and 38R; nonjudging of inner experience = 3R, 10R, 14R, 17R, 25R, 30R, 35R, and 39R; nonreactivity to inner experience = 4, 9, 19, 21, 24, 29, and 33. For the FFMQ subscales, scores can range from 8 to 40, except for non-reactivity to inner experience, which can range from 7 to 35. For the FFMQ subscales, higher scores represent higher subscale levels of mindfulness. Total scores are calculated by summing the subscale scores and range from 39-195, with higher scores indicating higher overall levels of mindfulness.
Change in rates of psychiatric diagnoses from baseline to 3 months | baseline and 3 months
  Change in rates of psychiatric diagnoses from baseline to 3 months will be measured using the Structured Clinical Interview for DSM-5 (SCID-5). The SCID-5 consists of a semistructured interview administered to participants by a clinician or trained mental health professional to determine participants' current and previous psychiatric diagnoses.

SECONDARY OUTCOMES:
Change in disinhibition from baseline to 8 weeks | baseline and 8 weeks
  Change in disinhibition from baseline to 8 weeks will be assessed by the Go/No-Go task (GNG). The GNG task is administered on the computer and asks participants to respond to visual stimuli that is presented continuously. Participants must make a motor response for the "go" stimulus and withhold a motor response for the "no-go" stimulus. The proportion of no-go targets in which an individual successfully withholds a motor response will provide a measure of response inhibition, with fewer errors indicating better response inhibition and a higher error rate indicating a greater tendency towards disinhibited behavior.
Change in disinhibition from 8 weeks to 3 months | 8 weeks and 3 months
  Change in disinhibition from 8 weeks to 3 months will be assessed by the Go/No-Go task (GNG). The GNG task is administered on the computer and asks participants to respond to visual stimuli that is presented continuously. Participants must make a motor response for the "go" stimulus and withhold a motor response for the "no-go" stimulus. The proportion of no-go targets in which an individual successfully withholds a motor response will provide a measure of response inhibition, with fewer errors indicating better response inhibition and a higher error rate indicating a greater tendency towards disinhibited behavior.
Change in attention from baseline to 8 weeks | baseline and 8 weeks
  Change in attention from baseline to 8 weeks will be assessed by the Stroop Color-Word Test. The Stroop Color-Word Test is a computerized task in which participants are required to name the color of a written color word while inhibiting the impulse to read the word itself. The difference between mean response times of correct responses on incongruent and control trials is used to compute an interference score, which provides a measure of attention, with lower scores indicating greater attentional deficits.
Change in attention from 8 weeks to 3 months | 8 weeks to 3 months
  Change in attention from 8 weeks to 3 months will be assessed by the Stroop Color-Word Test. The Stroop Color-Word Test is a computerized task in which participants are required to name the color of a written color word while inhibiting the impulse to read the word itself. The difference between mean response times of correct responses on incongruent and control trials is used to compute an interference score, which provides a measure of attention, with lower scores indicating greater attentional deficits.
Change in cognitive inflexibility from baseline to 8 weeks | baseline to 8 weeks
  Change in cognitive inflexibility from baseline to 8 weeks will be assessed by the Wisconsin Card Sorting Task (WCST). The WCST is a computerized task in which participants have to match a target card with one of four category cards under changing conditions. The number of incorrect responses that would have been correct for the preceding condition provides a measure of cognitive inflexibility, with higher scores indicating greater cognitive inflexibility.
Change in cognitive inflexibility from 8 weeks to 3 months | 8 weeks to 3 months
  Change in cognitive inflexibility from 8 weeks to 3 months will be assessed by the Wisconsin Card Sorting Task (WCST). The WCST is a computerized task in which participants have to match a target card with one of four category cards under changing conditions. The number of incorrect responses that would have been correct for the preceding condition provides a measure of cognitive inflexibility, with higher scores indicating greater cognitive inflexibility.
Change in emotion regulation from baseline to 8 weeks | baseline and 8 weeks
  Change in emotion regulation from baseline to 8 weeks will be measured using the 10-item Emotion Regulation Questionnaire (ERQ). The ERQ consists of two subscales, which are calculated by summing the following questions, which are scored 1-7 (none reverse scored): cognitive reappraisal = questions 1, 3, 5, 7, 8, and 10; expressive suppression = questions 2, 4, 6, and 9. For the ERQ subscales, scores can range from 1-42, with higher scores indicating higher use of that particular emotion regulation strategy and lower scores indicating less frequent use.
Change in emotion regulation from 8 weeks to 3 months | 8 weeks and 3 months
  Change in emotion regulation from 8 weeks to 3 months will be measured using the 10-item Emotion Regulation Questionnaire (ERQ). The ERQ consists of two subscales, which are calculated by summing the following questions, which are scored 1-7 (none reverse scored): cognitive reappraisal = questions 1, 3, 5, 7, 8, and 10; expressive suppression = questions 2, 4, 6, and 9. For the ERQ subscales, scores can range from 1-42, with higher scores indicating higher use of that particular emotion regulation strategy and lower scores indicating less frequent use.

OTHER OUTCOMES:
Participant satisfaction at 3 months | 3 months
  Participant satisfaction at 3 months will be measured quantitively with a 7-item Client Satisfaction Questionnaire (CSQ). Questions 1-3 on the CSQ assess participants' treatment satisfaction using a 10-point Likert scale. Questions 4-7 are opened-ended questions where participants can elaborate on their satisfaction with the treatment. Scores on questions 1-3 will be used to evaluate participant satisfaction and can range from 1-10. Total scores are calculated by summing the scores on questions 1-3 and can range from 3-30, with higher scores indicating greater participant satisfaction.
Participant satisfaction at 8 weeks | 8 weeks
  Participant satisfaction will be measured qualitatively with brief qualitative interviews performed at the end of the intervention, during which participants will have the opportunity to comment on their experiences in the group in an open-ended format. Responses during the interview will be recorded and evaluated using a thematic analysis.
Engagement (attendance) at 8 weeks | 8 weeks
  Engagement will be measured by session attendance rates. Attending 4 of the 8 group sessions is will be considered completion of the intervention and, thus, sufficient engagement.
Engagement (homework) at 8 weeks | 8 weeks
  Engagement will be assessed by the completion of daily homework as indicated by homework logs. Participants will be asked to practice mindfulness three days per week during the intervention period and will record the duration and type of meditation completed each day. Space will also be provided for participants to make note of anything they noticed about their practice. More frequent practice of mindfulness per week indicates higher levels of engagement.

CONTACTS AND LOCATIONS:
Overall Officials: Michele Levine, PhD, Principal Investigator — University of Pittsburgh Medical Center; Shannon Donofry, PhD, Principal Investigator — University of Pittsburgh-Psychology and (primarily) AHN Psychiatry & Behavioral Health Institute
Locations (1):
- Western Psychiatric Institute & Clinic, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
There are no plans and no requirements to share IPD.